CLINICAL TRIAL: NCT06784141
Title: Network-Based vs. Standardized Cognitive Behavioral Therapy in Chronic Primary Pain: A Single-Case Experimental Design With Randomized Baselines
Brief Title: Network-Based vs. Standardized Cognitive Behavioral Therapy in Chronic Primary Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Julia Glombiewski (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Julia Glombiewski, Clinical professor, Head of department clinical psychology and psychotherapy for adults, University of Kaiserslautern-Landau
Organization: University of Kaiserslautern-Landau (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POINT Pain 2
Record Dates: First submitted 2025-01-09; First posted 2025-01-20 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Chronic Primary Pain
Keywords: Chronic Pain; Single Case Experimental Design; Ecological Momentary Assessment; Network Analysis; Cognitive Behavior Therapy
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: The participants are assigned to one of the two possible intervention sequences: personalized CBT first and then standardized CBT, or in reverse order. In the personalized CBT, the participants will be allocated to one out of ten treatment modules according to their most relevant pain process. The same module will be used for the whole therapy phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- First standardized, second personalized CBT (Experimental): In this study arm, patients will first receive standardized and then personalized CBT. In the standardized CBT phase, a standardized CBT protocol will take place. In the personalized intervention phase, person-specific networks are estimated. A network-based algorithm indicates the treatment target. Participants will receive one out of ten CBT modules addressing their treatment target. A hybrid therapy option, i.e., partially online, will be available. The decision lies with the respective therapists and will be documented as a variable.
  Interventions: Behavioral: personalized Cognitive Behavior Therapy including third-wave; Behavioral: standardized Cognitive Behavior Therapy including third-wave
- First personalized, second standardized CBT (Experimental): In this study arm, patients will first receive standardized and then personalized CBT. In the personalized intervention phase, person-specific networks are estimated. A network-based algorithm indicates the treatment target. Participants will receive one out of ten CBT modules addressing their treatment target. In the standardized CBT phase, a manualized, standardized CBT will take place. A hybrid therapy option, i.e., partially online, will be available. The decision lies with the respective therapists and will be documented as a variable.
  Interventions: Behavioral: personalized Cognitive Behavior Therapy including third-wave; Behavioral: standardized Cognitive Behavior Therapy including third-wave

INTERVENTIONS:
Behavioral: personalized Cognitive Behavior Therapy including third-wave — In the personalized CBT, patients first complete 21 days of EMA with six assessment points daily to assess relevant processes of CPP models. Person-specific networks are estimated based on the EMA data. A network-based algorithm indicates the treatment target. The individual CBT modules are selected for the participants from a matching matrix that contains experts' module recommendations for specific treatment targets. After that, participants will receive one out of ten CBT modules addressing their treatment target. All treatment modules are based on evaluated treatment manuals and contain methods from Cognitive Behavior Therapy, Acceptance and Commitment Therapy or Mindful Selfcompassion.
Behavioral: standardized Cognitive Behavior Therapy including third-wave — The standardized CBT intervention is manual-based and contains five sessions of cognitive behavioral therapy. Based on the evaluated manual from EFFECT Back, a short version with 5 modules is used: attention control, relaxation techniques, behavioral activation, cognitive strategies, and consolidation.

SUMMARY:
Cognitive-behavioral therapy (CBT) has been shown to be an effective treatment for chronic primary pain (CPP), but overall effect sizes are small to moderate. Process orientation, personalization, and data-driven clinical decision-making may be able to address the heterogeneity among people with CPP and are thus promising ways to increase the effectiveness of CBT for CPP. In a previous study, the feasibility of personalized CBT for CPP using network analysis was investigated. Based on this work, the present study aims to compare this personalized CBT with a standardized CBT as treatment-as-usual condition.

In a balanced repeated measures design, a personalized CBT intervention is compared with a standardized CBT intervention. Participants are patients with CPP in German outpatient clinics. Primary and secondary outcome measures (disability, treatment expectations, pain intensity, working alliance, and side effects) will be collected after each study period. In addition, a SCED with randomized baselines will be embedded in the study, in which changes in processes relevant to chronic pain will be evaluated.

DETAILED DESCRIPTION:
Hypothesis:

Personalized CBT will achieve a comparable treatment effect to the standardized CBT condition, i.e. a stronger reduction in the outcome measures (intercept and slope).

Participants:

Recruitment takes place at selected university outpatient clinics throughout Germany. Patients will be recruited via the waiting list of the university's outpatient clinic, in cooperation with other currently running studies at the same university recruiting chronic pain patients, and via various media (e.g. newspaper articles) and doctors' offices. Study therapists will be recruited in the university's outpatient clinic as well. Inclusion criteria for patients are at least 18 years of age, having access to a smartphone, and the main diagnosis of chronic pain. The diagnosis will be checked using the brief version of the Diagnostic Interview for Mental Disorders (Mini-DIPS). For patients recruited via the waiting list, screening for suitability will take place during the first consultation at the university psychotherapy training center's outpatient clinic. Suitable participants will be informed about the study and referred if they agree to be contacted. Furthermore, patients that had to be excluded from other currently running studies will be referred if they agreed to be contacted as well.

Procedure & Measures:

Counterbalanced Repeated Measures Design: At this level, the primary outcome measure is pain disability index (PDI) and the WHO Disability Assessment Schedule 2.0 (WHODAS 2.0). Therapeutic alliance (Helping Alliance Questionnaire (HAQ), Working Alliance Inventory Short Revised (WAI-R); both therapist and patient version) and side effects (Negative Effects Questionnaire, NEQ) as well as expectations (Patient Questionnaire on Therapy Expectation and Evaluation, PATHEV) are collected as secondary outcome variables. These are collected before and after the diagnostic phase (A), after both interventions (C1, C2) and at follow-up (3 months). The HAQ, WAI-R, and NEQ constitute exceptions in this context. As these instruments pertain to the therapeutic relationship or the overall therapy process, they are not administered prior to the diagnostic phase, since no therapeutic contact has yet taken place. In addition, the therapist's case concept and a Perceived Causal Network (PECAN) of the therapist are collected after the diagnostic phase. Additional outcome measures are collected before the diagnostic phase (A), before the 3th baseline (B3) and at follow-up. As additional outcome measures the Depression Anxiety Stress Scale (DASS-21), the German Pain Solutions Questionnaire (PaSol), the Patient Global Impression of Change (PGIC) and Pain Self-Efficacy Questionnaire will be assed.

SCED: The participants begin with the standard diagnostic phase of routine clinical care (phase B, 5 sessions) with psychoeducation and the development of therapy goals. After a randomized baseline (phase A1, 1-3 weeks), the intervention phase (phase C) begins. Participants are randomly assigned to one of two groups. Group 1 begins with personalized CBT followed by standardized CBT whereas Group 2 begins with standardized CBT followed by personalized CBT. A second baseline takes place in both groups after the first intervention before the beginning of the second intervention (A2, randomized 1-3 weeks). After the two different therapeutic phases, another baseline (A3, 2 weeks) and afterwards an EMA phase of 3 weeks will be completed. In addition, there are two booster sessions with the therapist one and three months after the last therapy session. During the EMA phases, data will be collected 6 times per day. In all other phases, the questionnaires are asked 3 times a week.

Analysis:

To evaluate group differences, a multilevel analysis (MLM) is calculated to take the nested data structure into account. The effects within the individual participant are calculated at level 1 and across the participants at level 2. To determine the required sample size, we performed a data simulation assuming a normal distribution with two predictors in the MLM: Treatment and order of treatment. The simulation revealed that a sample size of 59 participants is required, with a power of 0.80 aimed for to detect small effect sizes. Based on the dropout rate observed in a previous pilot study, a sample size of N = 75 is planned.

The Bayes Factor and visual analysis are used to continuously evaluate the intervention effect at the individual level. In the visual analysis, we look at level, trend, variability, immediacy, overlap, and consistency.

ELIGIBILITY:
Inclusion Criteria:

* main diagnosis of chronic pain (i.e. pain persists for at least 6 months and is the most prominent/most burdensome symptom)
* subjective impairment/disability (yes-no)
* access to a smartphone compatible with the app mPath

Exclusion Criteria:

* acute hazard due to suicidality, substance abuse, and/or psychosis
* only migraine/headache or migraine/headache are the focus of pain
* analphabetism
* insufficient German knowledge
* current psychotherapy
* current participation in another intervention study
* physical inability to take part in therapy and study sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Pain Disability Index (PDI) | From baseline to posttest (an expected average of 22 weeks) to Follow-up-Assessment (an expected average of 6 month after posttest)
  The Pain Disability Index assesses the daily disability caused by pain in seven areas: family/domestic duties, recovery, social activities, work, sexuality, self-care, and life-sustaining activities. It has shown to be a valid instrument, displaying moderate test-retest reliability. Each item ranges from 0 to 10, with higher values indicating a greater disability due to pain.
WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | From baseline to posttest (an expected average of 22 weeks) to Follow-up-Assessment (an expected average of 6 month after posttest)
  A shorter version consisting of only twelve questions was developed based on the WHODAS 2.0. This abbreviated version also covers all six health domains, including two questions on a 5-point-scale per domain, with higher values indicating a greater disability due to pain.. During its development, it was demonstrated that the WHODAS 2.0 exhibits high internal consistency, strong test-retest reliability, and high validity in comparison with other instruments.

SECONDARY OUTCOMES:
Ecological Momentary Assessment questionnaire | from baseline to the end of the post-EMA (an expected average of 27 weeks)
  Throughout the whole study, the same questionnaire developed and in-evaluation for the use in Ecological Momentary Assessment will be applied. It assesses several therapy-relevant pain processes derived from common psychological models of chronic pain: catastrophizing, avoidance, depression (Fear-Avoidance model, Avoidance-Endurance model); thought suppression, task persistence, positive affect (Avoidance-Endurance model); acceptance, values (Psychological Flexibility); expectations (Predictive Coding); pain intensity, pain-related disability (Pain Experience); pain self-efficacy, self-compassion. The individual primary outcome will be the most relevant process for each participant according to the network from the first baseline. The items are rated on a scale from 0 to 10, with higher values indicating a worse outcome.
Working Alliance Inventory - Short Revised (WAI-SR) | From the end of the diagnostic phase to posttest (an expected average of 17 weeks) to Follow-up-Assessment (an expected average of 6 month after posttest)
  The WAI-SR measures the therapeutic alliance with three scales of four items each: attachment, agreement with the therapeutic approach, and therapeutic goals. There is a patient version (WAI-SR-P) and a therapist version (WAI-SR-T). The WAI-SR shows good reliability (α > 0.80) and convergent validity with the Helping Alliance Questionnaire (r > 0.64). The items are rated on a scale of 1 to 5, with higher values indicating a stronger therapeutic alliance.
Helping Alliance Questionaire (HAQ) | From the end of the diagnostic phase to posttest (an expected average of 17 weeks) to Follow-up-Assessment (an expected average of 6 month after posttest)
  The HAQ is a 12-item instrument designed to assess the therapeutic relationship and process variables. Total scores and two subscale scores on patient relationship satisfaction and success satisfaction can be calculated. The items are rated on a scale of 1 to 6, with higher scores indicating a stronger therapeutic alliance. It can be completed by both the patient and the therapist. The reliability and validity analyses showed satisfactory to good values in all areas.
Pain Intensity | From baseline to posttest (an expected average of 22 weeks) to Follow-up-Assessment (an expected average of 6 month after posttest)
  Pain Intensity will be measured on an 11-point numerical analogue scale over a period of 24 hours. The value 0 represents no pain, the maximum value 10 represents maximum possible pain.
Negative Effects Questionnaire (NEQ) | From the end of the diagnostic phase to posttest (an expected average of 17 weeks) to Follow-up-Assessment (an expected average of 6 month after posttest)
  The NEQ is an instrument for investigating negative effects in psychological treatments. The 20-item version of the NEQ shows comparable validity and reliability and uses a 5-point Likert-scale, with higher values indicating a stronger negative therapeutic effect.
Patient Questionnaire on Therapy Expectation and Evaluation (PATHEV) | From baseline to posttest (an expected average of 22 weeks) to Follow-up-Assessment (an expected average of 6 month after posttest)
  The PATHEV consists of three subscales: Hope of Improvement, Fear of Change, and Suitability. The reliability of the scales is good to sufficient. The questionnaire contains 11 items with a 5-point scale.

OTHER OUTCOMES:
German Pain Solutions Questionnaire (PaSol) | From baseline to posttest (an expected average of 22 weeks) to Follow-up-Assessment (an expected average of 6 month after posttest)
  The German version of the Pain Solutions Questionnaire assesses different coping strategies for pain with 14 items on a 7-point scale, with higher values indicating an improvement: solving pain, meaningfulness of life despite pain, acceptance of the insolubility of pain, and belief in a solution. It displays good reliability and validity and is sensistive for change.
Patient Global Impression of Change (PGIC) | From baseline to posttest (an expected average of 22 weeks) to Follow-up-Assessment (an expected average of 6 month after posttest)
  One item will be used to assess subjective treatment effects with the Patient Global Impression of Change. It will be answered on a 7-point scale, ranging from "no change" to "very much better".
Pain Self-Efficacy Questionnaire | From baseline to posttest (an expected average of 22 weeks) to Follow-up-Assessment (an expected average of 6 month after posttest)
  The Pain Self-Efficacy Questionnaire contains on 10 items using a 7-point scale, with higher values indicating an improvement. It was tested regarding comprehensibility and displays high reliability and validity. It also is sensitive to change.
Depression Anxiety Stress Scale (DASS-21) | From baseline to posttest (an expected average of 22 weeks) to Follow-up-Assessment (an expected average of 6 month after posttest)
  The DASS is a 42-item self report instrument and measures the three related negative emotional states of depression, anxiety and tension/stress and includes 7 items from each of the 3 subscales. The items are rated on a scale from 0 to 3, with higher values indicating stronger symptoms of depression, anxiety or stress. The internal consistency and concurrent validity were in acceptable to excellent ranges.

CONTACTS AND LOCATIONS:
Locations (1):
- RPTU Kaiserslautern-Landau, Klinische Psychologie und Psychotherapie des Erwachsenenalters, Landau, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hofmann VE, Glombiewski JA, Kininger F, Scholten S. How to personalise cognitive-behavioural therapy for chronic primary pain using network analysis: study protocol for a single-case experimental design with multiple baselines. BMJ Open. 2024 Dec 3;14(12):e089319. doi: 10.1136/bmjopen-2024-089319. PMID 39627123
- [Background] Vogt R, Haas J, Baumann L, Sander A, Klose C, Riecke J, Rief W, Bingel U, Maser D, Witthoft M, Kessler J, Zugaj MR, Ditzen B, Glombiewski JA. EFFects of Exposure and Cognitive behavioral Therapy for chronic BACK pain ("EFFECT-BACK"): study protocol for a randomized controlled trial. Trials. 2024 Mar 11;25(1):176. doi: 10.1186/s13063-024-08017-9. PMID 38468293
- [Background] Vogel F, Blanken TF, Burger J, Reichert J, Scholten S, Klintwall L. How perceived causal networks can complement case conceptualization, diagnostic classification, and data-based networks: An introduction to a method for constructing personalized networks. J Psychopathol Clin Sci. 2025 Oct;134(7):844-854. doi: 10.1037/abn0001036. Epub 2025 Aug 14. PMID 40811099
- [Background] Ustun TB, Chatterji S, Kostanjsek N, Rehm J, Kennedy C, Epping-Jordan J, Saxena S, von Korff M, Pull C; WHO/NIH Joint Project. Developing the World Health Organization Disability Assessment Schedule 2.0. Bull World Health Organ. 2010 Nov 1;88(11):815-23. doi: 10.2471/BLT.09.067231. Epub 2010 May 20. PMID 21076562
- [Background] Akerblom S, Perrin S, Rivano Fischer M, McCracken LM. Predictors and mediators of outcome in cognitive behavioral therapy for chronic pain: the contributions of psychological flexibility. J Behav Med. 2021 Feb;44(1):111-122. doi: 10.1007/s10865-020-00168-9. Epub 2020 Jul 8. PMID 32642875
- [Background] Williams ACC, Fisher E, Hearn L, Eccleston C. Psychological therapies for the management of chronic pain (excluding headache) in adults. Cochrane Database Syst Rev. 2020 Aug 12;8(8):CD007407. doi: 10.1002/14651858.CD007407.pub4. PMID 32794606
- [Background] Wright AGC, Woods WC. Personalized Models of Psychopathology. Annu Rev Clin Psychol. 2020 May 7;16:49-74. doi: 10.1146/annurev-clinpsy-102419-125032. Epub 2020 Feb 18. PMID 32070120
- [Background] Vlaeyen JWS, Crombez G. Behavioral Conceptualization and Treatment of Chronic Pain. Annu Rev Clin Psychol. 2020 May 7;16:187-212. doi: 10.1146/annurev-clinpsy-050718-095744. Epub 2019 Dec 10. PMID 31821023
- [Background] Wideman TH, Finan PH, Edwards RR, Quartana PJ, Buenaver LF, Haythornthwaite JA, Smith MT. Increased sensitivity to physical activity among individuals with knee osteoarthritis: relation to pain outcomes, psychological factors, and responses to quantitative sensory testing. Pain. 2014 Apr;155(4):703-711. doi: 10.1016/j.pain.2013.12.028. Epub 2013 Dec 28. PMID 24378879
- [Background] Beeckman M, Simons LE, Hughes S, Loeys T, Goubert L. A Network Analysis of Potential Antecedents and Consequences of Pain-Related Activity Avoidance and Activity Engagement in Adolescents. Pain Med. 2020 Feb 1;21(2):e89-e101. doi: 10.1093/pm/pnz211. PMID 31498397
- [Background] Liew BXW, Ford JJ, Briganti G, Hahne AJ. Understanding how individualised physiotherapy or advice altered different elements of disability for people with low back pain using network analysis. PLoS One. 2022 Feb 10;17(2):e0263574. doi: 10.1371/journal.pone.0263574. eCollection 2022. PMID 35143552
- [Background] Thompson EL, Broadbent J, Fuller-Tyszkiewicz M, Bertino MD, Staiger PK. A Network Analysis of the Links Between Chronic Pain Symptoms and Affective Disorder Symptoms. Int J Behav Med. 2019 Feb;26(1):59-68. doi: 10.1007/s12529-018-9754-8. PMID 30377989
- [Background] Borsboom D. A network theory of mental disorders. World Psychiatry. 2017 Feb;16(1):5-13. doi: 10.1002/wps.20375. PMID 28127906
- [Background] Anderson KO, Dowds BN, Pelletz RE, Edwards TW, Peeters-Asdourian C. Development and initial validation of a scale to measure self-efficacy beliefs in patients with chronic pain. Pain. 1995 Oct;63(1):77-83. doi: 10.1016/0304-3959(95)00021-J. PMID 8577493
- [Background] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Tait RC, Chibnall JT, Krause S. The Pain Disability Index: psychometric properties. Pain. 1990 Feb;40(2):171-182. doi: 10.1016/0304-3959(90)90068-O. PMID 2308763
- [Background] Mewes R, Rief W, Stenzel N, Glaesmer H, Martin A, Brahler E. What is "normal" disability? An investigation of disability in the general population. Pain. 2009 Mar;142(1-2):36-41. doi: 10.1016/j.pain.2008.11.007. Epub 2009 Jan 14. PMID 19147292
- [Background] Sielski R, Glombiewski JA, Rief W, Crombez G, Barke A. Cross-cultural adaptation of the German Pain Solutions Questionnaire: an instrument to measure assimilative and accommodative coping in response to chronic pain. J Pain Res. 2017 Jun 19;10:1437-1446. doi: 10.2147/JPR.S130016. eCollection 2017. PMID 28684921
- [Background] Germer CK, Neff KD. Self-compassion in clinical practice. J Clin Psychol. 2013 Aug;69(8):856-67. doi: 10.1002/jclp.22021. Epub 2013 Jun 17. PMID 23775511
- [Background] Rozental A, Kottorp A, Forsstrom D, Mansson K, Boettcher J, Andersson G, Furmark T, Carlbring P. The Negative Effects Questionnaire: psychometric properties of an instrument for assessing negative effects in psychological treatments. Behav Cogn Psychother. 2019 Sep;47(5):559-572. doi: 10.1017/S1352465819000018. Epub 2019 Mar 15. PMID 30871650
- [Background] Munder T, Wilmers F, Leonhart R, Linster HW, Barth J. Working Alliance Inventory-Short Revised (WAI-SR): psychometric properties in outpatients and inpatients. Clin Psychol Psychother. 2010 May-Jun;17(3):231-9. doi: 10.1002/cpp.658. PMID 20013760
- [Background] Guest G, Bunce A, & Johnson L. How many interviews are enough?: An experiment with data saturation and variability. Field Methods. 2006; 18(1): 59-82. https://doi.org/10.1177/1525822X05279903
- [Background] Morley S. Single-case methods in clinical psychology A practical guide (C. M., & C. J. M., Eds.). Routledge. 2018.
- [Background] Margraf J, Cwik JC, Suppiger A, & Schneider S. Mini-DIPS Open Access. Diagnostisches Interview bei psychischen Störungen [Short-Form of the Diagnostic Interview for Mental Disorders. Open Access]. 2017. https://www.kli.psy.ruhr-uni-bochum.de/dips-interv/klipsy/download/Mini-DIPS%20Open%20Access.pdf
- [Background] Green P, & MacLeod CJ. SIMR : an R package for power analysis of generalized linear mixed models by simulation. Methods in Ecology and Evolution. 2016; 7(4): 493-498. https://doi.org/10.1111/2041-210X.12504
- [Background] Nubling R, Kraft M, Henn J, Kriz D, Lutz W, Schmidt J, Wittmann W, Bassler M. [Testing the Psychometric Properties of the Helping Alliance Questionnaire (HAQ) in Different Health Care Settings]. Psychother Psychosom Med Psychol. 2017 Nov;67(11):465-476. doi: 10.1055/s-0043-111083. Epub 2017 Aug 30. German. PMID 28854445
- [Background] Schulte D. Messung der Therapieerwartung und Therapieevaluation von Patienten (PATHEV). Zeitschrift für Klinische Psychologie und Psychotherapie. 2005; 34(3): 176-187. https://doi.org/10.1026/1616-3443.34.3.176
- [Background] Mangels M, Schwarz S, Sohr G, Holme M, & Rief W. Der Fragebogen zur Erfassung der schmerzspezifischen Selbstwirksamkeit (FESS): Eine Adaptation des Pain Self-Efficacy Questionnaire für den deutschen Sprachraum. Diagnostica. 2009; 55(2): 84-93. https://doi.org/10.1026/0012-1924.55.2.84
- [Background] McCracken LM. Contextual cognitive-behavioral therapy for chronic pain. IASP Press. 2005.
- [Background] Nicholas M, Molloy A, Tonkin L, & Beeston L. Practical and positive ways of adapting to chronic pain Manage your pain. Souvenir press. 2003.
- [Background] Kleinstäuber M, Thomas P, Witthöft M, & Hiller W. Kognitive Verhaltenstherapie bei medizinisch unerklärten Körperbeschwerden und somatoformen Störungen (2. Aufl.). Springer. 2018.
- [Background] Germer CK, & Neff KD. Mindful Self-Compassion (MSC). In I. Itzvan (Ed.), The handbook of mindfulness-based programs: Every established intervention, from medicine to education. 2019;(357-367). Routledge.
- [Background] Main CJ, Keefe FJ, Jensen MP, Vlaeyen JWS, & Vowles KE. Fordyce's Behavioral Methods for Chronic Pain And Illness Republished with Invited Commentaries. IASP Press. 2015.
- [Background] de Vries RM, Morey RD. Bayesian hypothesis testing for single-subject designs. Psychol Methods. 2013 Jun;18(2):165-85. doi: 10.1037/a0031037. Epub 2013 Mar 4. PMID 23458719
- See also: Preregistration of the algorithmic decision-tool — https://doi.org/10.17605/OSF.IO/BNFWY
- See also: Preregistration of the EMA questionnaire development — https://doi.org/10.17605/OSF.IO/S4RMN
- See also: Preregistration of the feasibility study POINT Pain — https://clinicaltrials.gov/study/NCT06179784
- See also: Assessment app mPath — https://m-path.io/landing/